CLINICAL TRIAL: NCT05122117
Title: Impact of Photodynamic Therapy as an Adjunct to Non-surgical Periodontal Treatment on Clinical and Biochemical Parameters Among Patients Having Mild Rheumatoid Arthritis With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zohaib Akram (Other)
Responsible Party: Sponsor-Investigator, Zohaib Akram, Professor, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1234786
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis; Chronic Periodontitis
Keywords: photodynamic therapy; biomarkers; inflammation; Rheumatoid arthritis; chronic periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Periodontitis; Inflammation | interventions — Photochemotherapy; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue mediated photodynamic therapy (Experimental): Methylene blue (MB) with a concentration of 10 mg/mL was delivered inside the periodontal pocket. MB was injected inside in the selected periodontal pockets 4 - 6 mm with the help of a blunt needle and left for 1 min. Later, the periodontal pockets were flushed with distilled water for 3 min to remove the excess MB. The diode laser HELBO® TheraLite - Bredent Medical, Germany) of diameter 200 µm was used to deliver the light to initiate the disinfection process. Each participant underwent single session of laser exposure. The laser parameters such as wavelength, spot area, power output and laser energy were set at 660 nm, 0.028 cm2, 60 mW/cm2, and 150 mW, respectively. The laser was subjected for a period of 30 s in each pocket.
  Interventions: Device: Methylene blue mediated Photodynamic therapy; Procedure: Non-surgical periodontal therapy
- Scaling and root planing (Placebo Comparator): A single session of full-mouth ultrasonic scaling using a sterilized scaler was rendered to the control group. Deep pockets were additionally approached and cleaned by using manual 'After Fives' Gracey curette for root planning (Hu Friedy Gracey After Five Vision curette; HuFriedy, Chicago, USA). This session was followed by a polishing session. A motivational session was conducted where the patients were educated on the importance of maintaining a good oral hygiene by brushing their teeth twice daily followed by the regular use of dental floss and chlorhexidine mouth wash twice daily, respectively.
  Interventions: Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Device: Methylene blue mediated Photodynamic therapy — Methylene blue (MB) with a concentration of 10 mg/mL was delivered inside the periodontal pocket. MB was injected inside in the selected periodontal pockets 4 - 6 mm with the help of a blunt needle and left for 1 min. Later, the periodontal pockets were flushed with distilled water for 3 min to remove the excess MB. The diode laser HELBO® TheraLite - Bredent Medical, Germany) of diameter 200 µm was used to deliver the light to initiate the disinfection process. Each participant underwent single session of laser exposure. The laser parameters such as wavelength, spot area, power output and laser energy were set at 660 nm, 0.028 cm2, 60 mW/cm2, and 150 mW, respectively. The laser was subjected for a period of 30 s in each pocket.
  Other Names: Photodynamic therapy
  Arms: Methylene blue mediated photodynamic therapy
Procedure: Non-surgical periodontal therapy — A single session of full-mouth ultrasonic scaling using a sterilized scaler was rendered to the control group. Deep pockets were additionally approached and cleaned by using manual 'After Fives' Gracey curette for root planning (Hu Friedy Gracey After Five Vision curette; HuFriedy, Chicago, USA). This session was followed by a polishing session. A motivational session was conducted where the patients were educated on the importance of maintaining a good oral hygiene by brushing their teeth twice daily followed by the regular use of dental floss and chlorhexidine mouth wash twice daily, respectively.
  Other Names: Scaling and root planing

SUMMARY:
Purpose: To evaluate the efficacy of photodynamic therapy (PDT) as an adjunct to non-surgical periodontal therapy on the clinical periodontal and biochemical parameters among patients with rheumatoid arthritis (RA) having periodontitis.

Methods: A total of 50 RA patients with periodontitis were included. The subjects were equally divided into two groups: Group A - scaling and root planning (SRP) + PDT; Group B - SRP only, respectively. Plaque score (PS), bleeding on probing (BOP), pocket depth (PD) and clinical attachment level (CAL) were estimated. The biochemical parameters included the assessment of interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and rheumatoid factors (RFs). Multiple comparisons were established by employing the Bonferroni's post-hoc test for both clinical and laboratory biomarker data. The Mann-Whitney test was used to compute the p-value for intergroup comparisons. For intra-group comparisons, the p-value was computed with the help of Wilcoxon signed ranks test.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥25 years
* Satisfying the 2010 ACR/EULAR categorization criteria (with active RA with ≥6 joint involvement and under anti-RA medication ≥3 months)
* Patients having >20 teeth diagnosed with generalized (>30% of sites) chronic periodontitis with PD ≥ 4mm and/or CAL ≥ 4mm and vertical bone loss of at least 4 mm on radiography.

Exclusion Criteria:

* Patients who had underwent periodontal therapy or antimicrobial therapy in the last 6 months
* Any joint replacement
* Pregnancy/lactating mothers
* Patients having other forms of systemic diseases such as diabetes mellitus, hypertension or acquired immunodeficiency syndrome (AIDS)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Probing depth | 12 weeks
  Measurement of consecutive millimeter markings of the periodontal pocket depth
Clinical attachment level | 12 weeks
  Measurement of periodontal pocket depth along with recession

SECONDARY OUTCOMES:
Bleeding on probing | 12 weeks
  Presence or absence of bleeding indicated as '1' or '0', respectively
Plaque index | 12 weeks
  Presence or absence of plaque indicated as '1' or '0', respectively
Interleukin-6 | 12 weeks
  Assessment from gingival crevicular fluid
Tumor necrosis factor alpha | 12 weeks
  Assessment from gingival crevicular fluid

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia